CLINICAL TRIAL: NCT01730105
Title: Impact of Chronic Cold Exposure on Energy Metabolism in Humans
Brief Title: Chronic Cold Exposure and Energy Metabolism in Humans
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 130013; 13-DK-0013
Record Dates: First submitted 2012-11-17; First posted 2012-11-21 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2018-05-10

CONDITIONS: Healthy
Keywords: Adaptive Thermogenesis; Adipose Tissue; Body Composition; Body Weight Regulation; Brown Adipose Tissue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Background:

- Researchers are studying how metabolism and hormone levels change in response to mild changes in environmental temperature. Changes in metabolism may lessen with time because of hormonal adaptations. If this increase in metabolism continues for a longer period, mild cold exposure may cause weight loss. It is unclear whether exposure to a warmer temperature may cause opposite changes in metabolism. Researchers want to see if longer exposure (1 month) to different temperatures can affect how the body uses energy.

Objectives:

- To test changes in energy metabolism in response to different room temperatures.

Eligibility:

- Healthy men between 18 and 40 years of age.

Design:

* The entire study will last for 4 months. It will involve a screening visit and a 4-month inpatient stay at the National Institutes of Health Clinical Center. The inpatient stay will be in a private room at the Metabolic Clinical Research unit. Study participants will be required to stay in the Metabolic Clinical Research unit during the night, but are free to leave during the day.
* At the screening visit, participants will have a physical exam and medical history. Blood samples will be collected. A heart function test and diet questionnaire will also be given.
* During the first month, the temperature of the private room will be set at to 75.2 degrees F. This will allow the body to become used to the testing environment.
* During the second month, the temperature will be set to either a cool (66.2 degrees F) or a warm (80.6 degrees F) temperature.
* During the third month, the temperature will return to 75.2 degrees F.
* During the fourth month, the temperature will be altered to the opposite temperature to the one set in the second month.
* Throughout stay, participants will have daily temperature monitoring and will keep a food diary. Once a week, they will collect all of their urine for 24 hours. Once a month, they will spend 24 hours in a metabolic suite to study their metabolism rate.
* Throughout stay, the food will be provided as part of the study.
* During the first and third month (75.2 degrees F) the participants will be allowed to leave the Metabolic Clinical Research unit during the weekends, while during the second and forth month (66.2 or 80.6 degrees F), the participants will be allowed to spend one weekend out of the Metabolic Clinical Research unit.
* Other tests, such as body scans, fat tissue samples, and imaging studies, will be performed as needed.

DETAILED DESCRIPTION:
Obesity is a major health issue worldwide. Despite global research efforts, effective treatments for obesity are limited. There are two kinds of fat in the body: white fat and brown fat. White fat functions mainly as an energy-storing organ and in excess results in obesity and complications such as diabetes and high blood pressure. Brown fat on the other hand releases the energy stored in fat as heat. It protects small animals and newborn human infants from cold temperatures.

Recent advances in imaging techniques have revealed brown fat to be present in significant amount in adult humans. Using PET scanning, brown fat is shown to be more abundant in lean and younger individuals, suggesting that brown fat may regulate energy balance and metabolism. In a previous study we showed that following exposure to mild cold (19degree C/66degree F), the activity of brown fat was increased by nearly 10% and the energy expenditure by over 6%. Over time, these changes might result in substantial weight loss. However this has not been investigated and it is uncertain whether long-term cold exposure can sustain the increased activity of brown fat. In order to determine the therapeutic potential of brown fat activation, we designed a study investigating the effects of cold exposure over a long period.

We hypothesize that adult humans can be cold-acclimatized through mild cold exposure over a month. Brown fat activity can be increased and sustained by cold stimulation, which could result in beneficial metabolic changes in the body.

The aims of the current project are to:

1. determine whether brown fat can be stimulated by exposure to mild cold
2. investigate the metabolic consequences of long-term cold exposure

Volunteers will be randomly assigned to sleep overnight in the Metabolic Clinical Research Unit at NIH, set at either mild cold (19degree C/66degree F) or mild warm (27degree C/81degree F), with a lead-in period and a wash-out period before crossing over, during which the temperature will be ambient (24degree C/75 degree F). Volunteers can conduct their regular activities during the day. Each period will be 1 month in duration. At the end of each month, volunteers will be evaluated for their metabolic response to a mild cold challenge for 24 hours (19degree C/66degree F) to determine whether brown fat function and activity have been altered by temperature acclimatization in the previous month.

Significance: Based on its role in energy homeostasis and protection against obesity in animals, brown fat is likely to have a similar role in adult humans. Determining the contribution of brown fat-mediated cold acclimatization to long term energy balance may lead to novel treatment strategies of obesity.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Male
* Between 18-40 years old
* Willing to participate and provide informed consent

EXCLUSION CRITERIA:

* Hypo- or hyper-thyroid (history or TSH greater than 5.0 or less than 0.4 milli-international units per liter)
* Blood pressure greater than 140/90 millimeters of mercury (19) or current antihypertensive therapy
* History of cardiovascular disease
* BMI less than or equal to 20 or greater than or equal to 25 kilogram per cubic meter
* Diabetes mellitus or impaired fasting glycemia (fasting serum glucose greater than 100 grams per liter).
* Hypercholesterolemia (serum greater than or equal to 240 levels grams per liter), hypertriglyceridemia (plasma greater than or equal to 220 levels grams per liter) and/or use of antilipemic therapy.
* Liver disease or ALT serum level greater than two fold the upper laboratory reference limit.
* Iron deficiency (Ferritin less than 40 nanograms per milliliter males) (20).
* Renal insufficiency or estimated creatinine clearance less than 50 milliliter per minute (MDRD equation).
* Claustrophobia.
* History of illicit drug or alcohol abuse within the last 5 years; current use of drugs (by history) or alcohol (CAGE greater than 3).
* Psychiatric conditions or behavior that would be incompatible with safe and successful participation in this study
* Current use of medications/dietary supplements/alternative therapies known to alter thyroid function.
* Current use of antiplatelet or anticoagulants.
* Allergy to lidocaine.
* Current smoker or user of tobacco products
* Current participation in weight loss programs (dietary, exercise or pharmacological) or more than 3 kg weight changes in last 6 months
* Spending greater than 70% daily hours outdoors

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2012-11-17; Primary Completion 2014-06-24 (Actual); Study Completion 2018-05-10 (Actual)

PRIMARY OUTCOMES:
To determine the inducibility and plasticity of brown adipose tissue activity by chronic mild cold exposure in healthy adults.

SECONDARY OUTCOMES:
Evaluate the metabolic sequelae of chronic mild cold exposure
Evaluate the mechanisms underlying cold-induced metabolic changes

CONTACTS AND LOCATIONS:
Overall Officials: Kong Y Chen, Ph.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Ogden CL, Carroll MD, Kit BK, Flegal KM. Prevalence of obesity and trends in body mass index among US children and adolescents, 1999-2010. JAMA. 2012 Feb 1;307(5):483-90. doi: 10.1001/jama.2012.40. Epub 2012 Jan 17. PMID 22253364
- [Background] Cowburn G, Hillsdon M, Hankey CR. Obesity management by life-style strategies. Br Med Bull. 1997;53(2):389-408. doi: 10.1093/oxfordjournals.bmb.a011619. PMID 9246842
- [Background] Hankey CR. Session 3 (Joint with the British Dietetic Association): Management of obesity: Weight-loss interventions in the treatment of obesity. Proc Nutr Soc. 2010 Feb;69(1):34-8. doi: 10.1017/S0029665109991844. Epub 2009 Dec 15. PMID 20003637
- [Derived] Lee P, Smith S, Linderman J, Courville AB, Brychta RJ, Dieckmann W, Werner CD, Chen KY, Celi FS. Temperature-acclimated brown adipose tissue modulates insulin sensitivity in humans. Diabetes. 2014 Nov;63(11):3686-98. doi: 10.2337/db14-0513. Epub 2014 Jun 22. PMID 24954193